CLINICAL TRIAL: NCT05121493
Title: Study of Platelet Rich Plasma Drops to Moderate Clinically Significant Dry Eye
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, James V. Aquavella, MD, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004552
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet Poor Plasma Tear (Active Comparator)
  Interventions: Other: Platelet Poor Plasma Tear Drops
- Platelet Rich Plasma Tears (Experimental)
  Interventions: Other: Platelet Rich Plasma Tear Drops

INTERVENTIONS:
Other: Platelet Poor Plasma Tear Drops — Participant blood will be drawn and processed by the University of Rochester Transfusion Medicine and Blood Bank. Processing will isolate the platelet free fraction of the blood plasma. After processing, plasma should contain ≤ 5% concentration of white blood cells (WBC), red blood cells (RBC), and platelets when compared to the concentration before processing.
  Arms: Platelet Poor Plasma Tear
Other: Platelet Rich Plasma Tear Drops — Participant blood will be drawn and processed by the University of Rochester Transfusion Medicine and Blood Bank. Processing will isolate the platelet fraction of the blood plasma. After processing, plasma should contain ≤ 5% concentration of WBC and RBC and 100 x 10³ μl or ≥ 50% recovery of platelets when compared to the pre-platelet count.
  Arms: Platelet Rich Plasma Tears

SUMMARY:
This is a single center double-masked study with up to four visits. Subjects who have been diagnosed with dry-eye syndrome at Flaum Eye Institute will be enrolled. The purpose of the study is to determine if using platelet rich plasma drops can improve clinically significant dry eye in patients and determine if there is a difference with using two different uses of the plasma tear drops: platelet rich plasma tears and plasma tears without platelets.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be diagnosed with clinically significant dry eye.
* Subjects have no active ocular disease or allergic conjunctivitis.
* Subjects must not be using any topical ocular medications within two weeks prior to enrollment.
* Subjects must be willing and able to follow instructions.
* Subjects must have voluntarily agreed to participate in the study by signing the statement of informed consent.
* Subjects must meet plasma donor criteria as established by University of Rochester Transfusion Medicine & Blood Bank.

Exclusion Criteria:

* Is pregnant at the time of enrolment in the study determined by urine pregnancy test.
* Is currently on a course of antibiotics
* Is considered by the Investigator to not be a suitable candidate for participation and are not at risk for glaucoma.
* Is considered by the University of Rochester Transfusion Medicine & Blood Bank not a suitable candidate for blood donation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Mean change in acuity | baseline to 3 months
  Acuity will be measured using a Shack-Hartmann Wavefront Sensor. Subjects will be seated in front of the wavefront sensor. They will be asked to blink naturally fixate on the laser spot throughout the measurement protocol. While subjects fixate, the wavefront sensor delivers a brief flash of light to the subjects' retina. The light reflected out of the subjects' eye is collected to obtain measurements of wavefront aberrations of the eye. For optical quality assessments the measurements of wavefront aberrations will be acquired along the line-of-sight. The wavefront data acquired from the wavefront sensor will be described by Zernike coefficients, the most popular mathematical way to represent the ocular aberrations.
Mean change in breakup pattern to appear | baseline to 3 months
  This will be measured using a Placido Disk. The subject places their chin on a chin rest and look into the disk system. The system uses an incandescent or broad-band area LED for illumination.
Mean change in lipid coverage of the cornea with blinking | baseline to 3 months
  This will be measured using a Ellipsometer/Tearscope. This instrument uses a modified slit-lamp head restraint and an imaging system to visualize the surface of the subject's cornea. Structurally the system is a clinical slit-lamp system. However, the system uses an electronic camera instead of a human observer. The illumination system uses a diffuse ring illuminator instead of a slit-lamp. The data from this instrument identifies changes in the lipid thickness and the refractive index over the cornea.
Mean change in consistency of lipid compensation | baseline to 3 months
  This will be measured using a Ellipsometer/Tearscope. This instrument uses a modified slit-lamp head restraint and an imaging system to visualize the surface of the subject's cornea. Structurally the system is a clinical slit-lamp system. However, the system uses an electronic camera instead of a human observer. The illumination system uses a diffuse ring illuminator instead of a slit-lamp. The data from this instrument identifies changes in the lipid thickness and the refractive index over the cornea.
Mean change in temperature over the optical service | baseline to 3 months
  This will be measured using a Thermal Imaging System. A thermal imaging system will be used to provide spatially-resolved thermal maps of the subject's eyes and face adjacent to the eyes. This camera system is non-invasive and is mounted on a tripod about 12" from the subject's eyes. It images the heat that is emitted by the subject at frame rates from 2 to 10 Hz. The camera displays a spatially resolved map (approximately 0.2 x 0.2 mm pixel size) of the ocular surface temperature. IR detection is a convenient tool for instantaneous temperature measurement of the ocular surface and allows monitoring of time course change as well.

CONTACTS AND LOCATIONS:
Locations (1):
- Flaum Eye Institute at the University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No